CLINICAL TRIAL: NCT04270422
Title: Effect of Multidimensional Physiotherapy Based on Biopsychosocial Approach on Clinical Findings and Electroencephalography (EEG) Spectrum in Chronic Nonspecific Low Back Pain: A Randomized Controlled Trial
Brief Title: Effect of Multidimensional Physiotherapy in Chronic Nonspecific Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Iran University of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IranUMS
Record Dates: First submitted 2020-02-10; First posted 2020-02-17 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Low Back Pain, Mechanical
Keywords: Pain; Disability; Pain catastrophising; Quality of life; Fear of movement; Chronic non specific low back pain
MeSH Terms: conditions — Low Back Pain; Pain; Kinesiophobia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Multidimensional physiotherapy (Experimental): Multidimensional physiotherapy based on biopsychosocial, twice a week, 12 sessions
  Interventions: Other: Multidimensional physiotherapy
- Usual physiotherapy (Active Comparator): Usual evidence based physiotherapy, twice a week, 12 sessions
  Interventions: Other: Usual physiotherapy

INTERVENTIONS:
Other: Multidimensional physiotherapy — Multidimensional physiotherapy based on biopsychosocial approach
  Arms: Multidimensional physiotherapy
Other: Usual physiotherapy — Usual evidence based physiotherapy
  Arms: Usual physiotherapy

SUMMARY:
This study compares the effect of multidimensional physiotherapy to usual evidence-based physiotherapy in the treatment of chronic nonspecific low back pain in adults. Half of the participants will receive multidimensional physiotherapy based on biopsychosocial approach while the other half will receive usual evidence based physiotherapy.

DETAILED DESCRIPTION:
multidimensional physiotherapy treatment include: psychoeducation based on cognitive behavioral therapy (CBT), education, graded exposure, postural correction exercise, lifestyle change, and electrotherapy.

usual evidence-based physiotherapy include: electrotherapy, education, and trunk general exercises.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-50
* Low back pain for 3 months or more
* Disability based on Oswestry Disability Index (ODI) between 20-60
* Fear of movement based on Tampa scale of kinesiophobia >37
* Minimum level of education
* Native Persian speaking

Exclusion Criteria:

* Any evidence of e specific medical diagnosis
* Rheumatoid disease,fibromyalgia, neuropathy, progressive neurological disease
* History of headache, dizziness, nausea, epilepsy, migraines and mental disorder
* Beck's Anxiety Inventory> 26
* Beck's Depression Inventory II> 29
* Pregnancy
* Having other therapies during the present research

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2022-11-01 (Actual); Study Completion 2023-01-22 (Actual)

PRIMARY OUTCOMES:
Pain intensity(questionnaire): Numeric Rating Scale | At baseline
  Self reported pain intensity based on Numeric Rating Scale,that is composed of 0 (no pain at all) to 10 (worst imaginable pain).
Change of Pain intensity (questionnaire): Numeric Rating Scale | At 6 weeks, after 12 treatment sessions in 38 days
  Self reported pain intensity based on Numeric Rating Scale,that is composed of 0 (no pain at all) to 10 (worst imaginable pain).
Change of Pain intensity (questionnaire): Numeric Rating Scale | At 1 month
  Self reported pain intensity based on Numeric Rating Scale,that is composed of 0 (no pain at all) to 10 (worst imaginable pain).
Change of Pain intensity(questionnaire): Numeric Rating Scale | At 4 months
  Self reported pain intensity based on Numeric Rating Scale,that is composed of 0 (no pain at all) to 10 (worst imaginable pain).

SECONDARY OUTCOMES:
Quality of Life assessment | At baseline
  Self-reported quality of life based on health service (SF-36) questionnaire, the lower score the more disability and the higher score means the less disability.
Fear Avoidance Believes | At baseline
  Self reported Fear Avoidance Believes based on Fear Avoidance Believes questionnaire. A higher score indicates more strongly held fear avoidance beliefs.
Kinesiophobia | At baseline
  Self reported kinesiophobia based on Tampa scale of kinesiophobia. A higher score means more fear of movement.
Pain Catastrophizing | At baseline
  Self reported pain Catastrophizing based on Pain Catastrophizing Scale.The scale is a 13 item scale, with each item rated on a 5-point scale: 0 (Not at all) to 4 (all the time).
Disability | At baseline
  Self reported disability based on Oswestry disability scale Questionnaire. A higher number indicates a greater disability.
Forward flexion range of motion (ROM) | At baseline
  Forward flexion ROM measure by meter
Brain function | At baseline
  Relative power and absolute power of the frequency spectrum of EEG
Change in Quality of Life | At 6 weeks, after 12 treatment sessions in 38 days
  Self-reported quality of life based on health service (SF-36) questionnaire, the lower score the more disability and the higher score means the less disability.
Change of Fear Avoidance Believes | At 6 weeks, after 12 treatment sessions in 38 days
  Self reported Fear Avoidance Believes based on Fear Avoidance Believes questionnaire. A higher score indicates more strongly held fear avoidance beliefs.
Kinesiophobia | At 6 weeks, after 12 treatment sessions in 38 days
  Change of Self reported kinesiophobia based on Tampa scale of kinesiophobiaA higher score means more fear of movement.
Change of Pain Catastrophizing | At 6 weeks, after 12 treatment sessions in 38 days
  Self reported pain Catastrophizing based on Pain Catastrophizing Scale
Change of Disability | At 6 weeks, after 12 treatment sessions in 38 days
  Self reported disability based on Oswestry disability scale Questionnaire. A higher number indicates a greater disability.
Change of Forward flexion range of motion (ROM) | At 6 weeks, after 12 treatment sessions in 38 days
  Forward flexion ROM measure by meter
Change of Brain function | At 6 weeks, after 12 treatment sessions in 38 days
  Relative power and absolute power of the frequency spectrum of EEG
Change of Quality of Life | At 1 months
  Self-reported quality of life based on health service (SF-36) questionnaire, the lower score the more disability and the higher score means the less disability.
Change of Fear Avoidance Believes | At 1 months
  Self reported Fear Avoidance Believes based on Fear Avoidance Believes questionnaire. A higher score indicates more strongly held fear avoidance beliefs.
Change of Kinesiophobia | At 1 months
  Self reported kinesiophobia based on Tampa scale of kinesiophobiaA higher score means more fear of movement.
Change of Pain Catastrophizing | At 1 months
  Self reported pain Catastrophizing based on Pain Catastrophizing Scale.The scale is a 13 item scale, with each item rated on a 5-point scale: 0 (Not at all) to 4 (all the time).
Change of Disability | At 1 months
  Self reported disability based on Oswestry disability scale Questionnaire. A higher number indicates a greater disability.
Change of Forward flexion range of motion (ROM) | At 1 months
  Forward flexion ROM measure by meter
Change of Brain function | At 1 months
  Relative power and absolute power of the frequency spectrum of EEG
Change of Quality of Life | At 4 months
  Self-reported quality of life based on health service (SF-36) questionnaire, the lower score the more disability and the higher score means the less disability.
Change of Fear Avoidance Believes | At 4 months
  Self reported Fear Avoidance Believes based on Fear Avoidance Believes questionnaire.A higher score indicates more strongly held fear avoidance beliefs.
Change of Kinesiophobia | At 4 months
  Self reported kinesiophobia based on Tampa scale of kinesiophobiaA higher score means more fear of movement.
Change of Pain Catastrophizing | At 4 months
  Self reported pain Catastrophizing based on Pain Catastrophizing Scale.The scale is a 13 item scale, with each item rated on a 5-point scale: 0 (Not at all) to 4 (all the time).
Change of Disability | At 4 months
  Self reported disability based on Oswestry disability scale Questionnaire. A higher number indicates a greater disability.
Change of Forward flexion range of motion (ROM) | At 4 months
  Forward flexion ROM measure by meter
Change of Brain function | At 4 months
  Relative power and absolute power of the frequency spectrum of EEG

CONTACTS AND LOCATIONS:
Overall Officials: Javad Sarrafzadeh, Principal Investigator — IIran University of Medical Sciences
Locations (2):
- Iran (2):
  - Iran University of Medical Sciences, Tehran
  - School of Rehabilitation Sciences, Iran University of Medical Sciences, Tehran

IPD SHARING:
Plan to Share IPD: Yes
All data or results of the present study will present in an article that will be published after completing the study.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 8 months after completing the study
Access Criteria: Data access requests will be reviewed by the Corresponding Author will be required to sign a Data Access Agreement.

REFERENCES:
- [Derived] Bemani S, Sarrafzadeh J, Dehkordi SN, Talebian S, Salehi R, Zarei J. Effect of multidimensional physiotherapy on non-specific chronic low back pain: a randomized controlled trial. Adv Rheumatol. 2023 Dec 4;63(1):57. doi: 10.1186/s42358-023-00329-9. PMID 38049905
- [Derived] Bemani S, Dehkordi SN, Sarrafzadeh J, Talebian S, Salehi R, Zarei J. Efficacy of a multidimensional versus usual care physiotherapy on pain and electroencephalography (EEG) spectrum in chronic nonspecific low back pain: study protocol for a randomized controlled trial. Trials. 2021 Oct 7;22(1):679. doi: 10.1186/s13063-021-05580-3. PMID 34620205